CLINICAL TRIAL: NCT04795622
Title: Evaluation of the Effectiveness and Safety of the Ulthera® DeepSEE® System for Treating Skin Laxity in the Lower Face and Submentum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Collaborators: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M960101056
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Improvement in Skin Laxity of the Lower Face and Submentum
MeSH Terms: interventions — Treatment Delay

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Ulthera System (Experimental)
  Interventions: Device: Ultherapy treatment
- Delayed-treatment Ulthera System (Other)
  Interventions: Device: Untreated-control / delayed-treatment

INTERVENTIONS:
Device: Ultherapy treatment — Focused ultrasound energy delivered below the surface of the skin
  Arms: Treatment Ulthera System
Device: Untreated-control / delayed-treatment — Untreated-control, followed by Ultherapy treatment (focused ultrasound energy delivered below the surface of the skin)
  Arms: Delayed-treatment Ulthera System

SUMMARY:
1. Demonstrate superiority of treatment with the Ulthera DeepSEE System compared to untreated control for the improvement of skin laxity of the lower face and submental area.
2. Demonstrate the safety of treatment with the Ulthera DeepSEE System for the improvement of skin laxity of the lower face and submental area.

DETAILED DESCRIPTION:
Subjects in the study received a single treatment with Ulthera DeepSEE system on the midface, lower face, submental (under the chin) and upper neck area using 3 DeepSEE (DS) transducers (DS 10-1.5, DS 7-3.0, DS 7-4.5) at either Day 1 or Day 90. Subjects treated at Day 1 were followed for 180 days after treatment and subjects treated at Day 90 were followed for 90 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

- Mild to moderate lower face and/or submental laxity that is amenable to improvement with non-invasive intervention and is not severe enough for surgical intervention;

Exclusion Criteria:

* Scarring in area(s) to be treated;
* Any active implants (e.g., pacemakers or defibrillators) in the area(s) to be treated;
* Any metallic implants in area(s) to be treated;
* Any open wounds or lesions in the area(s) to be treated;
* Body mass index (BMI) less than 19 or greater than 30; or
* Gain or loss of ≥ 2 BMI units within the previous 90 days or has the intention to gain or lose ≥ 2 BMI units during the course of the trial.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (5):
- China (5):
  - Peking University First Hospital, Merz Investigational Site #0860003, Beijing
  - Air Force General Hospital, Merz Investigational Site #0860002, Beijing
  - Beijing Hospital, Plastic Surgery, Merz Investigational Site #0860029, Beijing
  - Shanghai 9th Hospital, Plastic Surgery, Merz Investigational Site #0860015, Shanghai
  - Huashan Hospital Shanghai, Merz Investigational Site #0860004, Shanghai

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 investigational sites in China.
Pre-assignment Details: Of the 213 screened subjects,12 were exited as screen failures and 201 subjects were enrolled and randomized in this study.
Groups:
- Treatment With Ulthera DeepSEE System: Subjects were randomized to receive a single treatment with Ulthera DeepSEE system at Day 1.
- Untreated Control/Delayed-treatment With Ulthera DeepSEE System: Subjects were randomized and were untreated until Day 90 and then received a single treatment with Ulthera DeepSEE system.
Period: Overall Study
Arm/Group | Treatment With Ulthera DeepSEE System | Untreated Control/Delayed-treatment With Ulthera DeepSEE System
Started | 101 | 100
Safety Evaluation Set (SES) | 97 | 96
Completed | 88 | 84
Not Completed | 13 | 16
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 2 | 3
Not completed — Other | 7 | 8

BASELINE CHARACTERISTICS:
Population: SES included all subjects who were treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Ulthera DeepSEE System | Untreated Control/Delayed-treatment With Ulthera DeepSEE System | Total
Number analyzed (Participants) | 97 | 96 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (7.57) | 47.3 (7.24) | 47.1 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 94 | 185
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 97 | 96 | 193

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Improvement in Lower Face and Submental Skin Laxity at Day 90
Description: Lower face and submental skin laxity were determined by three blinded evaluators after comparing Day 90 photographs with baseline photographs. Improvement was concluded if at least two evaluators assessed the Day 90 photographs as "improved" compared to baseline.
Time Frame: Day 90
Population: The full analysis set (FAS) included all subjects randomized with baseline photographs of acceptable quality.
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment With Ulthera DeepSEE System | Untreated Control/Delayed-treatment With Ulthera DeepSEE System
Number analyzed (Participants) | 96 | 100
percentage of subjects | 54.2 | 47.0
Statistical Analysis 1: Comparison: Treatment With Ulthera DeepSEE System vs Untreated Control/Delayed-treatment With Ulthera DeepSEE System; Test type: Superiority; Odds Ratio (OR) = 1.3545, 95% CI 2-sided [0.7530 to 2.4365]

2. Secondary Outcome: Displacement of Skin in the Submentum at Day 90
Description: Displacement of skin (in millimeters [mm]) in the submentum was determined by three-dimensional (3D) quantitative photographic analysis by comparing Day 90 photographs with baseline photographs. X-axis (lateral), Y-axis (vertical), and Z-axis (anterior to posterior) direction components were provided for both sides of the face combined (that is, overall).
Time Frame: Day 90
Population: FAS. Here "overall number of subjects analyzed" were subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Treatment With Ulthera DeepSEE System | Untreated Control/Delayed-treatment With Ulthera DeepSEE System
Number analyzed (Participants) | 92 | 96
millimeter (mm)
  X-axis | -0.0229 (0.5671) | 0.0571 (0.5125)
  Y-axis | -0.1693 (0.7151) | -0.1352 (0.6336)
  Z-axis | -0.2279 (1.1749) | -0.4086 (1.1509)
Statistical Analysis 1: Comparison: Treatment With Ulthera DeepSEE System vs Untreated Control/Delayed-treatment With Ulthera DeepSEE System; X-axis; Test type: Superiority; Point Estimate = -0.0856, 95% CI 2-sided [-0.2395 to 0.0683]
Statistical Analysis 2: Comparison: Treatment With Ulthera DeepSEE System vs Untreated Control/Delayed-treatment With Ulthera DeepSEE System; Y-axis; Test type: Superiority; Point Estimate = -0.0330, 95% CI 2-sided [-0.2268 to 0.1608]
Statistical Analysis 3: Comparison: Treatment With Ulthera DeepSEE System vs Untreated Control/Delayed-treatment With Ulthera DeepSEE System; Z-axis; Test type: Superiority; Point Estimate = 0.1791, 95% CI 2-sided [-0.1551 to 0.5133]

3. Secondary Outcome: Percentage of Subjects With Any Improvement on the Investigator Global Aesthetic Improvement Scale (iGAIS) at Day 90 as Assessed by the Treating Investigator in the Treatment Group
Description: iGAIS ratings (-3 to +3 scores; lower scores meant worse outcome) used baseline photographs for comparison. Improvement was defined as a rating of +1, +2, or +3 on the iGAIS.
Time Frame: Day 90
Population: FAS. This endpoint was pre-specified for the treatment group only.
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment With Ulthera DeepSEE System
Number analyzed (Participants) | 96
percentage of subjects | 96.8

4. Secondary Outcome: Percentage of Subjects With Any Improvement on the Subject Global Aesthetic Improvement Scale (sGAIS) at Day 90 as Assessed by the Subjects in the Treatment Group
Description: sGAIS ratings (-3 to +3 scores; lower scores meant worse outcome) used baseline photographs for comparison. Improvement was defined as a rating of +1, +2, or +3 on the sGAIS.
Time Frame: Day 90
Population: FAS. This endpoint was pre-specified for the treatment group only.
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment With Ulthera DeepSEE System
Number analyzed (Participants) | 96
percentage of subjects | 94.7

5. Secondary Outcome: Change From Baseline in FACE-Q Satisfaction With Lower Face and Jawline Score (Rasch-transformed) at Day 90, as Assessed by Subjects in Treatment Group
Description: The subject assessed satisfaction using the Face-Q Satisfaction with Lower Face and Jawline module (1 [very dissatisfied] to 4 [very satisfied] scores; Rasch transformed score 0-100; higher scores meant better outcome).
Time Frame: Baseline up to Day 90
Population: FAS. This endpoint was pre-specified for the treatment group only. Here "overall number of subjects analyzed" were subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With Ulthera DeepSEE System
Number analyzed (Participants) | 94
score on a scale | 30.3 (23.39)

6. Secondary Outcome: Number of Subjects With at Least One Treatment-related Treatment-emergent Adverse Events (TEAEs)
Time Frame: From first treatment (Day 1) up to end of the study (EOS) (Up to Day 180)
Population: SES.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment With Ulthera DeepSEE System: Subjects were randomized to receive a single treatment with Ulthera DeepSEE system at Day 1 and were followed for 180 days after treatment.
- Untreated Control/Delayed-treatment With Ulthera DeepSEE System: Subjects were randomized and were untreated until Day 90 and then received a single treatment with Ulthera DeepSEE system. Subjects were followed for 90 days after treatment.
Arm/Group | Treatment With Ulthera DeepSEE System | Untreated Control/Delayed-treatment With Ulthera DeepSEE System
Number analyzed (Participants) | 97 | 96
Participants | 36 | 34

ADVERSE EVENTS:
Time Frame: From first treatment (Day 1) up to end of the study (EOS) (Up to Day 180)
Description: SES. The investigator reported adverse events (AEs) systematically at each visit.
Arm/Group | Treatment With Ulthera DeepSEE System | Untreated Control/Delayed-treatment With Ulthera DeepSEE System
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/96
Serious Adverse Events (participants affected / at risk) | 3/97 | 0/96
Other Adverse Events (participants affected / at risk) | 34/97 | 32/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Ulthera DeepSEE System (N=97) | Untreated Control/Delayed-treatment With Ulthera DeepSEE System (N=96)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastric leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Ulthera DeepSEE System (N=97) | Untreated Control/Delayed-treatment With Ulthera DeepSEE System (N=96)
Application site pain (General disorders) | 22 | 24
Application site swelling (General disorders) | 16 | 3
Application site vesicles (General disorders) | 9 | 3
Application site erythema (General disorders) | 5 | 4
Application site discomfort (General disorders) | 6 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT04795622/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT04795622/SAP_001.pdf